CLINICAL TRIAL: NCT05964933
Title: Pulpotomy vs Root Canal Treatment for Teeth With Symptomatic Irreversible Pulpitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSRB 2023/00044
Record Dates: First submitted 2023-07-11; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-05

CONDITIONS: Pulpitis - Irreversible
Keywords: dental caries; deep caries; pulpotomy; root canal treatment; vital pulp therapy
MeSH Terms: conditions — Dental Caries | interventions — Pulpectomy

STUDY DESIGN:
Intervention Model Description: Study subject (tooth) will be randomized in a 1:1 allocation ratio between the two treatment groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be done to the outcomes assessors to reduce bias during radiographic healing assessment. Participants also will not be informed of which treatment they are undergoing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Pulpotomy (Active Comparator): The tooth will be treated with Complete Pulpotomy.
  Interventions: Procedure: Complete Pulpotomy
- Pulpectomy and Root Canal Treatment (Active Comparator): The tooth will be treated with Pulpectomy and Root Canal Treatment.
  Interventions: Procedure: Pulpectomy and Root Canal Treatment

INTERVENTIONS:
Procedure: Complete Pulpotomy — Complete caries removal and excision of the entire coronal pulp to the level of the root canal orifices will be performed. After haemostasis, the pulp chamber will be filled with Biodentine® and a final direct restoration placed in 1 or 2 visits.
  If there is no bleeding from the exposed pulp, pulpectomy and root canal treatment will be performed instead, and the patient will be excluded from the study.
  Other Names: Full Pulpotomy; Coronal Pulpotomy
  Arms: Complete Pulpotomy
Procedure: Pulpectomy and Root Canal Treatment — After complete caries removal and pulp exposure, Pulpectomy will be performed to remove all pulp tissues. Conventional root canal treatment will be performed using rotary instrumentation followed by obturation with gutta percha and traditional sealers in 1 or 2 visits. A final restoration will be placed to ensure a good coronal seal, and this may include full coronal coverage restorations if clinically indicated.
  Other Names: Conventional Root Canal Treatment; Non-surgical Endodontic Treatment
  Arms: Pulpectomy and Root Canal Treatment

SUMMARY:
This study is a randomised controlled trial for complete pulpotomy as an alternative to root canal treatment for teeth with clinical diagnosis of symptomatic irreversible pulpitis (i.e. signs and symptoms indicative of irreversible pulpitis) conducted at the National University Centre for Oral Health Singapore (NUCOHS) Endodontic unit. Up to 70 teeth, 35 in each group, will be enrolled.

Clinical and radiographic outcome data will be collected and analysed, and a parallel cost-effectiveness analysis will also be undertaken to examine the potential costs and benefits of pulpotomy. A process evaluation will also be conducted to assess the acceptability of the intervention to both dentists and patients, while exploring the barriers and enablers to implementation.

DETAILED DESCRIPTION:
Mature permanent teeth with deep caries/restorations and symptoms indicative of irreversible pulpitis (moderate to severe spontaneous lingering pain) will be included in the study. The teeth will be randomised to receive one of two treatments: RCT or complete pulpotomy (n=35 in each group).

Baseline clinical and radiographic data will be collected at the first visit. In addition, patients (or their guardians, if relevant) will be invited to complete the acceptability and willingness to pay questionnaires for health economics analysis at both the first visit and at 12 months from the date of completed treatment. Pain data will be collected via a pain diary after completion of treatment at days 3 and 7 post-treatment. Patients will be clinically and radiographically reviewed at 6 and 12 months from the date of completed treatment. Review clinical data collected will include the absence of pain (and details on the nature of pain, if relevant), tenderness to percussion and palpation, presence of a swelling or a sinus tract, pathological mobility, structural integrity of tooth, intact and non-defective restoration, and response to electric pulp testing (for the pulpotomy group only). Radiographic data collected will include the presence of periapical radiolucency, presence of inter-radicular radiolucency, presence of resorption, and presence of calcifications. The need for any further intervention (including details of any procedure) or any adverse events or unscheduled visits over the follow-up period will also be recorded.

Success will be defined as 1) the absence of pain indicative of irreversible pulpitis, 2) the absence of signs and symptoms indicative of acute or chronic periapical disease, and 3) the absence of radiographic evidence of failure including radiolucency or resorption. SPSS Statistical Package (IBM SPSS Statistics) will be used for all statistical analysis, with the significance level for all statistical tests set at p-value<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or older
* Mature permanent tooth with deep caries/restorations
* Symptoms indicative of irreversible pulpitis (moderate to severe spontaneous lingering pain)
* Tooth is responsive to cold and electric pulp test (EPT) sensibility testing
* Tooth is restorable and can be adequately isolated during treatment
* One tooth (molar or premolar) per patient.

Exclusion Criteria:

* Teeth with active periodontal disease (pocket depth >5mm)
* Teeth indicated for elective root canal treatment for restorative purposes
* Teeth with apical periodontitis
* Patients with complex medical histories that may affect their caries experience and healing ability (immunocompromised, radiotherapy etc.)
* Patients who are unable to consent
* History of trauma to the tooth
* Presence of apical radiolucency
* Patients who are pregnant or breast-feeding
* Teeth with any evidence of purulence or excessive bleeding that cannot be controlled with a cotton pellet with 2-4% hypochlorite for 10 minutes

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Composite measure is defined by the change from baseline pain and radiographic status at 6 months and again at 12 months. | 6, 12 months
  Composite measure defined as:
  1. absence of pain indicative of irreversible pulpitis;
  2. absence of signs and symptoms indicative of acute or chronic periapical disease;
  3. absence of radiographic evidence of failure including radiolucency or resorption.

SECONDARY OUTCOMES:
Numeric Rate Scale (NRS): minimum value = 0 (best outcome), maximum value = 10 (worst outcome) | 3, 7 days
  A patient reported outcome of pain experienced and use of analgesia in the immediate post-operative period, collected through a Numeric Rating Scale (NRS).
Restoration: the restoration remains intact and adapts completely to the prepared cavity margins. | 6, 12 months
  The presence of a structurally integral tooth with an intact, non-defective restoration.
A "yes" or "no" response when the Cold Test and Electric Pulp Test are applied on the treated tooth. | 6, 12 months
  Positive sensibility response on electrical pulp test (EPT) for the Pulpotomy group only.
N5. Clinicians examine the treated tooth to determine if there is pathology that resulted from the treatment. | 12 months
  Absence of need for any further intervention during the follow-up period or any adverse event.
Data to be collected include time spent on receiving the treatment, cost of treatment, and patients' willingness to pay for treatment. | 12 months
  A parallel process evaluation and health economics analysis will be completed using data collected from participants at baseline and at 12 months.
Radiographic appearance of the dental pulp and its canal(s) at baseline will be compared to that at 12 months. | 12, months
  Radiographic evidence of pulp calcification in response to Pulpotomy (applicable to the Pulpotomy group only).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, PhD, Principal Investigator — National University Hosptial, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No